CLINICAL TRIAL: NCT06821945
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Design, Exploratory Clinical Trial to Evaluate the Safety and Efficacy of Olanzapine Titration Schedule in Patients With Schizophrenia
Brief Title: A Clinical Trial to Evaluate the Safety and Efficacy of Olanzapine Titration Schedule in Patients With Schizophrenia
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: BR-OLZ-CT-201
Record Dates: First submitted 2025-02-06; First posted 2025-02-12 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gradual titration group (Experimental)
  Interventions: Drug: BR5402A; Drug: BR5402B; Drug: BR5402C; Drug: BR5402C-1; Drug: BR5402D; Drug: BR5402D-1
- Conventional titration group (Active Comparator)
  Interventions: Drug: BR5402A-1; Drug: BR5402B-1; Drug: BR5402C; Drug: BR5402C-1; Drug: BR5402D

INTERVENTIONS:
Drug: BR5402A — Subjects take the investigational products once a day
  Arms: Gradual titration group
Drug: BR5402A-1 — Subjects take the investigational products once a day
  Other Names: Placebo of BR5402A
  Arms: Conventional titration group
Drug: BR5402B — Subjects take the investigational products once a day
  Arms: Gradual titration group
Drug: BR5402B-1 — Subjects take the investigational products once a day
  Other Names: Placebo of BR5402B
  Arms: Conventional titration group
Drug: BR5402C — Subjects take the investigational products once a day
Drug: BR5402C-1 — Subjects take the investigational products once a day
  Other Names: Placebo of BR5402C
Drug: BR5402D — Subjects take the investigational products once a day
Drug: BR5402D-1 — Subjects take the investigational products once a day
  Other Names: Placebo of BR5402D
  Arms: Gradual titration group

SUMMARY:
The objective of this clinical trial is to evaluate the safety and efficacy of olanzapine titration schedule in patients with schizophrenia

ELIGIBILITY:
Inclusion Criteria:

* Of patients with schizophrenia in accordance with DSM(Diagnostic and Statistical Manual of Mental Disorders)-5 diagnostic criteria, who are judged that administration of low dose is more appropriate than initial recommended dose or standard titration dose of olanzapine to consider medical conditions by investigator
* Patients with the duration of schizophrenia for more than 1 year at screening visit(Visit 1)

Exclusion Criteria:

* Patients diagnosed schizophrenia spectrum and other psychotic disorder(e.g. schizoaffective disorder, etc.), bipolar disorder, depressive disorder, etc., in accordance with DSM(Diagnostic and Statistical Manual of Mental Disorders)-5 diagnostic criteria at screening visit(Visit 1)
* Patients with a history of hospitalization for worsening schizophrenia within 12 weeks at screening visit(Visit 1)

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-05-30 (Actual); Primary Completion 2027-05 (Estimated); Study Completion 2027-05 (Estimated)

PRIMARY OUTCOMES:
The mean change of PANSS(Positive and Negative Syndrome Scale) total score | 1, 2, 3, 5, 9 weeks from baseline(Visit 2)
Incidence of treatment-emergent adverse events | From the administration of investigational products prescribed at baseline(Visit 2) to 11 weeks(Visit 8)

CONTACTS AND LOCATIONS:
Locations (2):
- South Korea (2):
  - Kyungbook National university hospital, Daegu
  - Hanyang University Guri Hospital, Guri-si

IPD SHARING:
Plan to Share IPD: No